CLINICAL TRIAL: NCT06493851
Title: The Effect of Hyperbaric Oxygen Therapy (HBOT) for Acceleration Recovery After Anterior Cruciate Ligament Reconstruction (ACLR): a Prospective, Randomized Control Study.
Brief Title: The Effect of Hyperbaric Oxygen Therapy for Acceleration Recovery After Anterior Cruciate Ligament Reconstruction(ACLR)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 166-23
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-07

CONDITIONS: Anterior Cruciate Ligament Reconstruction
Keywords: hyperbaric oxygen therapy
MeSH Terms: interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Intervention Model Description: hyperbaric oxygen therapy (2ATA, 100% oxygen) vs. sham (1.2ATA, 21% oxygen)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- hyperbaric oxygen therapy (HBOT) active treatment (Active Comparator): The HBOT protocol consists of 6 weeks protocol including 5 daily HBOT sessions per week (total of 30), each session lasts 90 minutes, of 100% oxygen at 2 atmosphere absolute (ATA) with 5-minute air breaks every 20 minutes.
  Interventions: Device: hyperbaric oxygen therapy
- hyperbaric oxygen therapy (HBOT) Sham treatment (Sham Comparator): The sham HBOT protocol consists of 6 weeks protocol including 5 daily sham HBOT sessions per week (total of 30), each session includes breathing 21% oxygen by mask in a sham multiplace chamber. Sham pressure will go up to 1.2 ATA during the first five minutes of the session (to stimulate the pressure sensation in the ears), and then decrease during the next 5 minutes to 1.03 ATA for 90 minutes with 5-minute air breaks every 20 minutes.
  Interventions: Device: hyperbaric oxygen therapy

INTERVENTIONS:
Device: hyperbaric oxygen therapy — The HBOT protocol consists of 6 weeks protocol including 5 daily HBOT sessions per week (total of 30), each session lasts 90 minutes, of 100% oxygen at 2 atmosphere absolute (ATA) with 5-minute air breaks every 20 minutes.
  Investigational product:
  Multiplace hyperbaric oxygen chamber (Haux Starmed 2700, Germany) located at the Sagol center for hyperbaric medicine and research, Shamir (Assaf-Harofeh) Medical Center, Israel.

SUMMARY:
The aim of the current study is to evaluate the effect of HBOT for acceleration recovery after ACLR.

DETAILED DESCRIPTION:
ACL rapture (Anterior cruciate ligament reconstruction rehabilitation) is a common injury in sports and cause severe functional problem. The big concern with this injury is the time to return to sport, this is the interest of the athlete.

The preferred treatment today when it comes to active athletes is to have an anterior cruciate ligament reconstruction (ACLR) ,the return to high function and sports after anterior cruciate ligament reconstruction (ACLR) surgery lasts about 8 months.

In the last few years, knowledge has been accumulating regarding the effectiveness of the new hyperbaric oxygen protocols in accelerating the healing of wounds and tissue damage. it was found that Hyperbaric oxygen therapy (HBOT) for ligament injuries in mice improves the quality and speed of recovery. The effect of HBOT on the rate of ligament healing has not yet been properly tested in humans.

The constant search for accelerated recovery in sports injuries along with the benefit of the HBOT in tissue healing processes encouraged the need to investigate the rate of recovery after a sports injury under HBOT. Two previous human studies in which medial collateral tear was tested showed positive effect on pain, physical outcome (decreased edema, range of motion and maximal knee flex) and accelerate the return to play. These findings with the fact that ACL injuries are common among athletes and can limit return to sports, reinforce the need to examine the effect of HBOT following ACLR in the terms of improving and speeding up recovery.

The aim of the current study is to evaluate the effect of HBOT for acceleration recovery after ACLR.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects willing and able to read, understand and sign an informed consent
2. Age 18-45
3. Anterior cruciate ligament tear for reconstruction (with or without meniscal repair).

Exclusion Criteria:

1. Inability to attend scheduled clinic visits and/or comply with the study protocol
2. Additional injury
3. An inability to perform MRI.
4. Active malignancy
5. Chest pathology incompatible with pressure changes (including active asthma)
6. Ear or sinus pathology incompatible with pressure changes
7. History of epilepsy
8. Claustrophobia
9. Previous knee surgery
10. Participation in another study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-15 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
International Knee Documentation Committee | Change from Baseline immediately after the intervention
  The aim of the international knee documentation committee (IKDC) is to detect improvement or deterioration in symptoms, function, and sport activity following knee impairment. Scores range from 0 points (lowest level of function or highest level of symptoms) to 100 points (highest level of function and lowest level of symptoms).

SECONDARY OUTCOMES:
Knee MRI | Change from Baseline immediately after the intervention
  At each of the evaluations, patients will undergo structural MRI scanning. Images will be acquired on MAGNETOM Vida 3T Scanner, configured with a channel receiver knee coils (Siemens Healthcare, Erlangen, Germany) at Shamir medical centre.
  Edema and haemorrhage are seen as increased signal in the substance of the ACL in an acute injury.
Laxity ligament test | Change from Baseline immediately after the intervention
  Laxity ligament test includes 2 parts: 1- Lachman, anterior drawer, pivot - Manual assessment of the knee joint stabilization, The result will recorded as normal to severely abnormal according to criteria established by the IKDC. 2- KT-1000 - The KT-1000 test is knee arthrometer assessment for ACL laxity, The results of the KT-1000 examination will be recorded as normal to severely abnormal according to guidelines established by the IKDC .
physical measurement - ROM | Change from Baseline immediately after the intervention
  ROM - Range of motion will be assessed with the patient in the supine position using a goniometer, passive knee flexion will be rated normal to severely abnormal according to established IKDC guidelines.
physical measurement - Edema | Change from Baseline immediately after the intervention
  Edema- One of the common measurement methods in research is knee perimetry, the assessor measures the knee girth at 3 points: the fold at the popliteal fossa (P0), 5 cm above P0 (PA), and 5 cm below P0 (PB). Data on perimetry were calculate.
physical measurement - Vas for pain | Change from Baseline immediately after the intervention
  Vas for pain - Pain scales are useful for the assessment of postoperative pain and based on self-reporting and represent subjective pain intensity, The evaluation is performed according to the IKDC : Scores range from 0 points (lowest level of function or highest level of symptoms) to 100 points (highest level of function and lowest level of symptoms).
physical measurement - Maximal quadriceps power by dynamometer | Change from Baseline immediately after the intervention
  Maximal quadriceps power by dynamometer - Quadriceps strength after ACLR usually assessed by isometric dynamometry and comparison the strength of the ACLR limb with the uninjured limb.
Functional scores- (PROM) | Change from Baseline immediately after the intervention
  Tegner Lysholm knee scoring scale - patient-reported outcome measure (PROM) ,The total score is the sum of each response to the eight questions and may range from 0-100. Higher scores indicate a better outcome with fewer symptoms or disabilities, Score are categorized as excellent (95-100), good (84-94), fair (65-83), and poor (<64).
Functional scores - Vas for global rating of knee function | Change from Baseline immediately after the intervention
  Vas for global rating of knee function - measure the participation restrictions experienced during activities of daily living and sports by patients with a history of ACLR. rating of function by assessing the level of knee function on a 0 to 100 scale, with 0 points representing complete loss of function due to their knee injury and 100 points representing their level of function prior to their knee injury.
Short form health survey (sf-36) | Change from Baseline immediately after the intervention
  Quality of life questionnaire, scale of 0-100, higher score means better outcome
Functional measurement | Change from Baseline immediately after the intervention
  Balance Error Scoring System (BESS) - minimally clinical important difference (MCID) is 3 points and MDC intra-rater 7.3 points.
Functional measurement - (SEBT) | Change from Baseline immediately after the intervention
  Modified Star Excursion Balance Test (SEBT) - Minimally clinical important difference (MCID) is 3.5% difference between the two legs.
Functional measurement - Single Hop test | Change from Baseline immediately after the intervention
  Single Hop test - MDC- score improved by 21.98 for women and 21.81 for man (as a % of leg length).

CONTACTS AND LOCATIONS:
Overall Officials: Shai a Efrati, MD, Principal Investigator — Asaf-Harofhe MC
Locations (1):
- The Sagol Center for Hyperbaric Medicine and Research Shamir Medical Center (Assaf Harofeh), Zrifin, Israel

IPD SHARING:
Plan to Share IPD: No